CLINICAL TRIAL: NCT03773406
Title: Timing of Transcranial Direct Current Stimulation (tDCS) Combined With Speech and Language Therapy (SLT): An Intervention Development Study for Aphasia
Brief Title: Timing of Transcranial Direct Current Stimulation (tDCS) Combined With Speech and Language Therapy (SLT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leora Cherney, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90IFRE0020
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Aphasia
Keywords: Aphasia, tDCS, Script training, Functional language, Naming
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Offline tDCS-before therapy (Active Comparator): Participants will receive 20 minutes of tDCS prior to the 40 minute speech-language therapy session.
  Interventions: Device: Offline tDCS-before therapy
- Offline tDCS-after therapy (Active Comparator): Participants will receive 20 minutes of tDCS after the 40 minute speech-language therapy session.
  Interventions: Device: Offline tDCS-after therapy
- Online tDCS (Active Comparator): tDCS will be applied at the beginning of the 40 minute speech-language therapy session and will last for 20 minutes.
  Interventions: Device: Online tDCS
- Sham tDCS (Sham Comparator): Sham tDCS will be applied at the beginning of the 40 minute speech-language therapy session.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Offline tDCS-before therapy — Direct current stimulation will be delivered using a battery-driven constant current stimulator. 2mA of direct current will be applied for 20 minutes to the angular gyrus region of the brain. We will use a standard-of-care treatment - script training - to provide speech-language therapy to our subjects. The scripting treatment will be delivered by a computer program that provides script training in an interactive conversational context.
  Arms: Offline tDCS-before therapy
Device: Sham tDCS — Stimulation will be given for a total 30 seconds (including ramp-up and ramp-down of current) and then the tDCS device will be turned off. The brief stimulation will produce tDCS-induced sensation so that participants will not be aware when the tDCS was turned off .We will use standard-of-care treatment - script training - to provide speech-language therapy to our subjects. The scripting treatment will be delivered by a computer program that provides script training in an interactive conversational context.
  Arms: Sham tDCS
Device: Offline tDCS-after therapy — Direct current stimulation will be delivered using a battery-driven constant current stimulator. 2mA of direct current will be applied for 20 minutes to the angular gyrus region of the brain. We will use a standard-of-care treatment - script training - to provide speech-language therapy to our subjects. The scripting treatment will be delivered by a computer program that provides script training in an interactive conversational context.
  Arms: Offline tDCS-after therapy
Device: Online tDCS — Direct current stimulation will be delivered using a battery-driven constant current stimulator. 2mA of direct current will be applied for 20 minutes to the angular gyrus region of the brain. We will use a standard-of-care treatment - script training - to provide speech-language therapy to our subjects. The scripting treatment will be delivered by a computer program that provides script training in an interactive conversational context.
  Arms: Online tDCS

SUMMARY:
Aphasia is an acquired (typically left-hemisphere) multi-modality disturbance of language that impacts around 2 million people in the USA. Aphasia impacts language production and comprehension as well as reading and writing. The ramifications of aphasia extend beyond language impairment to negatively impacting a person's social, vocational, and recreational activities. Currently, the most effective way to treat aphasia is with speech-language therapy (SLT). However, even if SLT is intensive, persons with aphasia are left with residual language delays. Recent research suggests that pairing SLT with transcranial direct current stimulation (tDCS) a non-invasive, safe, low-cost form of brain stimulation may aid language recovery in persons with aphasia. However, results from tDCS studies are inconclusive. The success of tDCS in combination with SLT could depend on the timing of tDCS since tDCS-induced effects depend on the neuronal state of the brain-networks at the time of the stimulation. In this study, the differential impact of tDCS before behavioral SLT (offline-before therapy), tDCS after SLT (offline-after therapy), and tDCS concurrently with SLT (online) on functional language recovery in persons with aphasia will be investigated. Sham tDCS (i.e., SLT alone) as a control group will also be included in the study. The investigators hypothesize that both offline and online tDCS will improve language functioning than sham tDCS.

DETAILED DESCRIPTION:
tDCS Implementation:

2mA of direct current for 20 minutes will be delivered using a constant current stimulator via two electrodes in saline soaked sponges. To stimulate the left angular gyrus, a cathodal electrode inside a saline soaked sponge (5 x 3cm) will be placed over the CP5 according to the 10-20 international system for EEG electrode placement. The electrodes will be secured in position by a custom-built EEG cap that will be marked with the location for angular gyrus. The investigators will then confirm that the cathodal electrode is over the left angular through the use of neuronavigation. The "return" anode electrode will be placed in a saline soaked sponge (5 x 5cm) on the center of the supraorbital region.

At the beginning of the tDCS, current will slowly ram-up during the first few seconds until it reaches 2mA. The ramp-up process will acclimate the participants to tDCS-induced sensations (e.g., itching). At the end of the tDCS sessions, current will slowly ramp down in the last few seconds to 0mA. The total duration of the 2mA current will be maintained for 20 minutes. For sham stimulation, the investigators will place the electrodes in the same location as the real tDCS groups with stimulation ending after few seconds. The brief stimulation will produce tDCS-induced sensations so that participants will not be aware when the tDCS stopped delivering direct current

Speech-Language Treatment:

Standard-of-care treatment - script training will be used to provide SLT to our participants. The treatment will be delivered via a computer program, Aphasia Scripts ®, whereby a virtual therapist interactively guides the participants through treatment steps. Scripts will be five to ten sentences and developed from common templates about topics relevant to daily life (e.g., asking questions at the grocery store, ordering in a restaurant). The advantage of using a computer program instead of a human therapist is that it removes extraneous variables associated with human therapists (e.g., different levels of encouragement) and this, together with the use of script templates, ensures treatment fidelity across participants.

Duration of an individual subject's participation in the study:

Subjects will be requested to come for baseline sessions (3 to 4 hours) before the actual experiment. The baseline assessments may be done over two visits. In the baseline session the subjects' aphasia severity will be assessed. The participants will also perform baseline tasks of language and cognition in this session. Subjects will then participate in 3 weeks of tDCS and SLT (i.e., 15 sessions). The sessions will consist of 40 minutes of SLT and 20 minutes of tDCS. Subjects will be asked to return for an assessment immediately following the end of treatment and for follow-up testing after 4 and 8 weeks. Therefore, total number of visits will be 19-23 sessions (depending on how many visits are needed for the assessments) over a period of three months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with diagnosis of fluent or non-fluent aphasia subsequent to a left-hemisphere infarct(s) that is confirmed by a MRI or CT scan
* Aphasia quotient on the WAB of 35-85
* At least 6 months post onset of aphasia (this is beyond the stage of spontaneous recovery)
* 18- 80 years of age
* Premorbidly fluent in English
* Premorbidly right-hand dominant per the Edinburg Handedness Inventory
* Visual acuity of 20/40 corrected
* Auditory acuity no worse than 30 dB HL on pure tone testing, aided in the better ear.
* Education greater than 12th grade

Exclusion Criteria:

* Any other neurological condition (other than cerebral vascular disease) that could impact language and cognition such as Alzheimer's disease, Parkinson's disease, primary progressive aphasia, and traumatic brain injury
* Active substance use
* Individuals with epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in trained conversational script. | 3 weeks.
  Changes in accuracy and rate of production on a trained conversational script from pre to post-treatment.

SECONDARY OUTCOMES:
Change in untrained conversational script | 3 weeks
  Changes in accuracy and rate of production on an untrained conversational script from pre to post-treatment.
Change in the Aphasia Quotient (AQ) of Western Aphasia Battery-Revised (WAB-R) | 3 weeks
  Changes in WAB-R AQ from pre and post treatment.
Maintenance of trained conversational script | 7 weeks
  Accuracy and rate of production of trained conversational script at 4 weeks post-treatment
Maintenance of trained conversational script | 11 weeks
  Accuracy and rate of production of trained conversational script at 8 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leora Cherney, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ashaie SA, Engel S, Cherney LR. Timing of transcranial direct current stimulation (tDCS) combined with speech and language therapy (SLT) for aphasia: study protocol for a randomized controlled trial. Trials. 2022 Aug 17;23(1):668. doi: 10.1186/s13063-022-06627-9. PMID 35978374